CLINICAL TRIAL: NCT04369274
Title: A Repeated Measures Trial of Temporary Automated Manual Ventilation Versus Noninvasive Oxygenation or Conventional Ventilation for the Treatment of COVID-19 ARDS
Brief Title: Repeated Measures Trial of Temporary Automated Manual Ventilation Versus Noninvasive Oxygenation or Conventional Vent
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The epidemic of Covid pneumonia requiring large scale mechanical ventilation has abated and the need to explore alternate ventilatory devices has resolved.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Keith Marill, Emergency Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P001051
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilator
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiration, Artificial

STUDY DESIGN:
Intervention Model Description: The design is a case series with repeated measures analysis. All patients will receive the experimental treatment as well as conventional ventilation and unassisted oxygenation as observed prior to initiation of mechanical ventilation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Interventional (Experimental): All subjects will briefly be placed on the automated BVM compressor device. Measurements obtained while on this device will be compared to those obtained in the same subject prior to mechanical ventilation and while on a conventional ventilator.
  Interventions: Device: Mechanical ventilation with the automated BVM compressor

INTERVENTIONS:
Device: Mechanical ventilation with the automated BVM compressor — Mechanical ventilation is accomplished with a device that mechanically squeezes a manual bag valve instead of by hand. The rate and volume of compression are adjustable, and the device has appropriate alarms and safety features.

SUMMARY:
The COVID-19 pandemic has led to a potential shortage of life-saving mechanical ventilators. The purpose of this study is to determine whether a novel simpler to device, the automated bag-valve-mask (BVM) compressor, can be used to provide assisted ventilation temporarily to patients in need. This includes patients with COVID-19 lung infection and respiratory failure. If successful, this would increase the pool of total available ventilator hours to alleviate any shortage.

DETAILED DESCRIPTION:
This study will be performed in the emergency department and ICU's of Massachusetts General Hospital (MGH). Thirty patients requiring mechanical ventilation will be enrolled. The design is a case series with repeated measures analysis. All patients will receive the experimental treatment as well as conventional ventilation and unassisted oxygenation as observed prior to initiation of mechanical ventilation. The compressor used will be manufactured by Spiro LLC / 10xbeta based on the open source MIT design. The device is powered by an uninterrupted power supply from a standard electrical outlet and it alarms if unplugged.

The patient will be moved into a negative pressure room. After patients with respiratory failure are intubated and stabilized on a conventional ventilator, they will receive 15 minutes of artificial respirations with the automated compressor with the conventional ventilator standing by. They will be returned to the conventional respirator after this period, or sooner if necessary. The endotracheal tube will be briefly clamped during the rapid transition from one device to another to minimize aerosolization of any viral particles and to retain any PEEP.

If the initial study period demonstrates successful respiratory support, then the procedure may be repeated once with doubling of the automated compressor treatment time to 30 minutes. There will be a minimum 15-minute observation period with conventional mechanical ventilation between the two study periods. Additionally, there will be one hour of data collection after the study periods. The total duration of the two intervention periods, the intervening period and data collection is two hours. The primary outcome is arterial oxygenation.

Patients are chemically paralyzed to facilitate intubation as part of standard care. Rocuronium is typically used for intubating chemical paralysis in the MGH emergency department. It has a half-life of 66 minutes. A single repeat bolus will be provided if needed to ensure chemical paralysis for the duration of the study. If the patient is already intubated and no longer chemically paralyzed, than one bolus of rocuronium, and a second as needed, or just a temporary increase in ongoing sedation will be provided to minimize spontaneous respiration. The airway circuit will be continuously monitored with a separate pressure and flow monitor (Nico) with recorded digital output throughout the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Patient may be diagnosed with Covid-19 based on clinical presentation and available laboratory studies including specific Covid-19 testing.
* Patient with imminent respiratory failure or status post respiratory failure receiving mechanical ventilation, or requiring mechanical ventilation for airway protection or other cause.
* Evidence of no pulmonary disease, or mild to moderate ARDS based on:

  * fraction of inspired oxygen (FiO2) ≤ 60% with arterial oxygen saturation > 90%
  * positive end expiratory pressure (PEEP) ≤ 12 cm H20
* Using an adaptive trial design, the first 10 patients must require mechanical ventilation for reasons other than COVID-19 infection such as airway protection due to overdose, seizure, stroke, or trauma. The next 10 patients may have COVID-19 infection, but must demonstrate lung compliance ≥ 40 ml/cm H2O. If these 10 patients demonstrate a satisfactory course associated with treatment, then the final 10 patients may have lung compliance ≥ 30 ml/cm H2O. Satisfactory treatment course will include, at a minimum: oxygen saturation > 90%, with PEEP ≤ 12 cm H2O.

Exclusion Criteria:

* Lack of informed consent from patient, if deemed having capacity, or from surrogate if not
* Too medically unstable to participate in study per treating clinician
* Patients requiring more than one vasopressor medication for blood pressure support
* Age > 65 years
* Clinical evidence of acute coronary syndrome (ACS) including angina, or ECG evidence of acute ischemia or dysrhythmia
* Chronic lung disease including chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, or pulmonary hypertension
* Gross laboratory abnormalities including, when available: liver function tests (LFT) > 5x normal, C-reactive protein (CRP) > 200 mg/L, ferritin > 2000 µg/L, creatine phosphokinase (CPK) > 3x normal, D-Dimer > 2500 ng/ml
* Previously enrolled subject
* Children
* Pregnant women
* Estimated body mass index (BMI) greater than 30
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Arterial oxygenation | Measurement 10 minutes after onset of initial period of automatic compressed ventilations
  Arterial oxygenation obtained as measured by noninvasive pulse oximetry and arterial blood gas.
Arterial oxygenation | Measurement 20 minutes after onset of second period of automatic compressed ventilations
  Arterial oxygenation obtained as measured by noninvasive pulse oximetry and arterial blood gas.

SECONDARY OUTCOMES:
Expired pressure of carbon dioxide. | 2 hour total study period.
  Expired carbon dioxide (CO2) pressure will be measured continuously with a monitor in the airway circuit.
Airway pressure | 2 hour total study period.
  The pressure (cm H2O) of inspired and expired air in the airway circuit while the subject is mechanically ventilated will be measured continuously using a Nico monitor.
Heart rate | 2 hour total study period.
  Subject heart rate (beats per minute) will be measured continuously using a telemetry monitor,
Blood pressure | 2 hour total study period.
  Subject blood pressure (mm Hg) will be measured episodically every 5 minutes using an automated arm cuff.
Airway flow | 2 hour total study period.
  The flow (L/min) of inspired and expired air in the airway circuit while the subject is mechanically ventilated will be measured continuously using a Nico monitor.

OTHER OUTCOMES:
Mortality | Duration of hospitalization, up to 2 months
  The subject will be followed clinically to assess for recovery and survival or death.

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Marill, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Husseini AM, Lee HJ, Negrete J, Powelson S, Servi AT, Slocum AH, Saukkonen J. Design and Prototyping of a Low-Cost Portable Mechanical Ventilator. J Med Device. 2010 Jun 1;4(2):027514. doi: 10.1115/1.3442790. Epub 2010 Aug 9. PMID 32328214